CLINICAL TRIAL: NCT03147222
Title: Hip Fracture Caregiver Intervention - Function Focused Care: Fracture Care at Home
Brief Title: Function Focused Care: Fracture Care at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ann Gruber-Baldini, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00072220; 1R21AG054143-01 (NIH)
Record Dates: First submitted 2017-05-03; First posted 2017-05-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Fractures, Bone; Dementia
Keywords: fragility fracture; dementia; intervention
MeSH Terms: conditions — Fractures, Bone; Dementia

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fracture Care at Home (Experimental): A trained FFC coach will visit each caregiver and fracture participant in the home for a 1-2 hour session once a week for 8 weeks.
  Interventions: Behavioral: Fracture Care at Home

INTERVENTIONS:
Behavioral: Fracture Care at Home — This is a graduated, functionally-based intervention, paired with caregiver interactions for enhancing functional abilities. Caregivers are encouraged to have the fracture participant actively participate in their own activities of daily living and incorporate functional activities into daily routines. An intervention coach will discuss care related challenges with the caregiver to identify dependency problems, motivate the caregiver to help foster independence in the care recipient, and provide guidance in addressing behavioral symptoms associated with cognitive limitation that may occur during caregiving. The coach is guided by interventions designed by PTs, OTs, and a nurse practitioner expert in FFC. The intervention includes 1) initial assessment of participant, caregiver, and environment, 2) coaching and mentoring of caregivers regarding use of effective motivational strategies, 3) goal setting, and 4) on-going motivation and evaluation.
  Other Names: Function Focused Care (FFC) for the Cognitively Impaired

SUMMARY:
This pilot study will evaluate the feasibility of implementing an intervention in the home setting that is specifically designed to coach and mentor caregivers as they assist individuals with Alzheimer's disease and related dementia (ADRD) who have fractured a hip to perform everyday activities and engage in more physical activity.

DETAILED DESCRIPTION:
Prior research by the Baltimore Hip Studies (BHS) has shown that it is possible to improve function, increase physical activity, and improve behavioral symptoms among long term care residents with ADRD and to effectively coach and mentor caregivers through a care practice, Function Focused Care for the Cognitively Impaired (FFC-CI), that focuses on having caregivers teach, cue, model, and assist cognitively impaired individuals to perform functional tasks and engage in physical activity, while minimizing behavioral symptoms. This study will determine if a revised intervention, Function Focused Care for the Cognitively Impaired: Hip Care at Home (aka, Hip Care at Home), can be implemented in a home setting.

The Hip Care at Home intervention will include an initial evaluation of the hip fracture participant, caregiver, and home setting by an interdisciplinary care team including a physical therapist (PT), occupational therapist (OT), and a coach (nurse or nurse's aide) trained in the function focused care (FFC) approach. The FFC coach will then work with the primary informal (family or friend, unpaid) caregiver to integrate the recommended environmental, behavioral, and physical interventions into the home setting, with weekly visits.

ELIGIBILITY:
FRACTURE PARTICIPANTS

Inclusion Criteria:

* Fragility fracture (hip, spine, femur/thigh, wrist, humerus/arm)
* Pre-fracture diagnosis of Alzheimer's disease or related dementia from chart, informant, or through AD8 score of 2+
* Age 65+ at time of fracture
* Completed usual rehabilitation
* Discharged to the community after rehabilitation ends (i.e., private home or assisted living)
* Availability of a caregiver (i.e., family relative or non-relative, unpaid, informal) providing ADL or IADL care or oversight at least weekly

Exclusion Criteria:

* Pathologic fracture
* Not community-dwelling (e.g., nursing home resident) prior to fracture
* Bedbound during the 6 months prior to fracture
* No caregiver or caregiver refuses study participation
* Study clinician thinks participant is not a good candidate for study

Not returning to the community before one year after fracture (can go to assisted living)

CAREGIVER PARTICIPANTS

Inclusion Criteria:

* Identified as a caregiver (i.e., family relative or non-relative, unpaid, informal) who will help or supervise the fracture participant with ADL or IADL tasks after discharge from rehab
* Helping or supervising thefracture participant with one or more ADL or IADL tasks at least weekly when screened for this study OR plans to be the primary person providing care at least weekly after the fracture participant is discharged from rehab

Exclusion Criteria:

* Not English speaking
* Living more than 40 miles from the hip fracture participant
* Unable to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | 8 weeks
  Data regarding feasibility will include numbers of participants contacted, enrolled, drop-outs/withdrawals, and completing intervention, adverse events, and total time to implement intervention.
Treatment Fidelity | 8 weeks
  Treatment fidelity of the intervention will include recording of adherence and logs of intervention tasks and problems by the interdisciplinary care team and FFC coach regarding barriers to implementation of the intervention and open-ended interviews with caregivers about their experiences with the intervention.

SECONDARY OUTCOMES:
Physical Activities of Daily Living (PADLs) - fracture participant outcome | 8 weeks
  Physical activities of daily living (PADLs) assess the fracture participant's receipt of assistance in 15 PADLs with an instrument whose structure is similar to Jette's Functional Status Index and incorporates activities from the Older Americans Resources and Services (OARS) Instrument PADL scale and those used by Cummings et al.
Instrumental Activities of Daily Living (IADLs) - fracture participant outcome | 8 weeks
  Instrumental activities of daily living (IADLs) are measured by 7 items from the OARS.
Short Physical Performance Battery (SPPB) - fracture participant outcome | 8 weeks
  Short Physical Performance Battery (SPPB) will be used to assess timed physical performance of balance, gait, strength, and endurance. Walking speed over 3 meters and a single timed chair rise without using arms will also be assessed.
MotionWatch to Monitor Physical Movement - fracture participant outcome | 8 weeks
  A MotionWatch manufactured by CamNtech Ltd., a compact, lightweight, body-worn activity monitoring device, will be placed on the wrist of the fracture participant at each measurement interview (baseline and follow-up) and removed 5 days later by study personnel. The MotionWatch is intended to monitor limb or body movements during daily living and sleep and may be used to document physical movement associated with applications in physiological monitoring.
Modified Mini-Mental State Examination (3MS) - fracture participant outcome | 8 weeks
  Global cognition will be assessed using the Modified Mini-Mental State Examination (3MS), which also be used to describe severity of ADRD. This measure will be used to describe the extent of the cognitive impairment in people with ADRD in the sample and selecting a comparison group from existing data.
Neuropsychiatric Inventory (NPI) - fracture participant outcome | 8 weeks
  Behavioral and affective outcomes will examine the impact on caregiver rated behavioral symptoms of ADRD using the Neuropsychiatric Inventory (NPI), which includes items on 10 behavioral disturbances: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, and aberrant motor activity. These are all rated by the caregiver.
Cornell Scale for Depression in Dementia (CSDD) - fracture participant outcome | 8 weeks
  The Cornell Scale for Depression in Dementia (CSDD) was specifically developed to assess signs and symptoms of major depression in patients with dementia. Caregivers will be interviewed on each of the 19 items on the scale and instructed to base her/his report on observations of the fracture participant's behavior during the week prior to the interview.
Adverse Events | 8 weeks
  Falls and other adverse events, including hospitalization, nursing home placement, and death will be recorded throughout the study.
Improvement in Knowledge of FFC - caregiver outcome | 2 weeks and 8 weeks after the start of the intervention
  Knowledge of FFC will be assessed using the Knowledge of Function and Behavior Focused Care Activities Test after the information is presented and again at end of study.
Self-Efficacy for Functional and Physical Activities - caregiver outcome | 8 weeks
  Self-Efficacy for Functional and Physical Activities is a 10-question survey to the caregiver about their confidence in their ability to encourage the hip fracture participant to undertake difference activities of daily living independently. Responses are either 'Yes' or 'No'.
Outcomes Expectations for Function and Physical Activity - caregiver outcome | 8 weeks
  Outcomes Expectations for Function and Physical Activity is a 9-item survey given to caregivers about the extent to which they agree that with statements about caregiving and care recipient independence.
Improvement in Performance of FFC - caregiver outcome | 3 weeks and 6 weeks after the start of the intervention
  Performance of FFC care will be assessed using the Function Focused Care Behavior Checklist. Observations will be done by the FFC coach in the home setting as part of the regular weekly intervention visits at 3 weeks and 6 weeks after the start of intervention. Immediate feedback will be provided to the caregiver following the observed care interactions (e.g., positive reinforcement for function focused care will be provided or information about missed opportunities for function focused care to be provided) and the FFC coach will work toward immediate increased integration of the recommended interventions during routine care.
Zarit Burden Interview - caregiver outcome | 8 weeks
  Caregiver burden will be assessed using the Zarit Burden Interview, a 22-item scale answered by caregivers, response options ranging from 0 (Never) to 4 (Nearly Always). Factors capture personal strain and role strain.
Center for Epidemiologic Studies Depression Scale (CES-D) - caregiver outcome | 8 weeks
  Caregiver depressive symptoms will be measured using the 20-item version of the Center for Epidemiologic Studies Depression Scale (CES-D). Possible scores range from 0-60.
Falls Efficacy Scale International (FES-I) | 8 weeks
  The Falls Efficacy Scale International (FES-I) will be used to assess fear of falling in fracture participants and fear of falling in caregivers for themselves and their care recipients.

OTHER OUTCOMES:
Assessment of Environment for Impact on Physical Activity | 3 weeks and 6 weeks after the start of the intervention
  Assessment of Environment for Impact on Physical Activity is a visual checklist indicating whether the described environmental component is present or absent. This measure will be included at baseline to tailor the intervention, but will be repeated at follow-up as a potential intermediate outcome. Environment assessments will be done by the FFC coach and recommendations for change discussed with caregiver and initiated as approved. Additionally, changing the environment to optimize function and physical activity (e.g., providing access to open areas for walking, pleasant destinations, and rest areas along pathways) will also facilitate the integration of the Hip Care at Home intervention.
Goal Attainment | 3 weeks and 6 weeks after the start of the intervention
  Knowledge from the environment, caregiver beliefs/culture of the home environment, and the Physical Capability Assessment will be used to set goals. Up to four fracture participant goals are listed on the Goal Attainment Scale and then scored on their progress where scores can range from -8 to 8 with score of 0 indicating expected progress and positive score indicates greater than expected progress. This measure will be included at baseline to tailor the intervention, but will be repeated at follow-up as a potential intermediate outcome.
Care Goal Identification | 3 weeks and 6 weeks after the start of the intervention
  The Care Goal Identification Form is a 3 part form used to identify problems, goals to address those problems, and ways to incorporate technology into the solutions. This measure will be included at baseline to tailor the intervention, but will be repeated at follow-up as a potential intermediate outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gruber-Baldini, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No